CLINICAL TRIAL: NCT04431050
Title: Evaluation of a Single Use Point of Care Device for the Diagnosis of Influenza and Other Respiratory Pathogens in Clinical Upper Airway Samples Using Isothermal Amplification - a Feasibility Study
Brief Title: Evaluation of a Single Use Point of Care Device for the Diagnosis of Respiratory Pathogens
Acronym: SIMPLIFI
Status: Terminated | Type: Observational
Why Stopped: Terminated due to covid-19- not reinstated due to low flu admissions
Sponsor: Imperial College London (Other)
Collaborators: Sense Biodetection Limited (Unknown)
Responsible Party: Sponsor
Other Study IDs: 19SM5486
Record Dates: First submitted 2020-02-24; First posted 2020-06-16 (Actual); Results first posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Human Influenza; Respiratory Syncytial Virus Infections; Rhinoviral Infections; Enterovirus Infections; Metapneumovirus Infection; Parainfluenzae Viral Infections
MeSH Terms: conditions — Influenza, Human; Respiratory Syncytial Virus Infections; Enterovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — One nasal swab taken from each participant for diagnostics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected influenza or other respiratory viral infection.: Any adult presenting to the Accident & Emergency department with influenza like illness or a febrile illness associated with symptoms such as cough, sore throat or rhinorrhoea, and for whom a respiratory viral screen is clinically indicated.
  For the purposes of this study one nasal swab will be taken from consenting adults.
  Interventions: Diagnostic Test: Point of care testing of respiratory viruses.

INTERVENTIONS:
Diagnostic Test: Point of care testing of respiratory viruses. — Single use point of care diagnostic device.

SUMMARY:
This study evaluates a single use point of care diagnostic test in the diagnosis of influenza and other respiratory viral infections in adults. Participants will have a sample taken from their nose using a swab. The swab will be gently mixed in a liquid solution which will then be transferred into the device for testing.

DETAILED DESCRIPTION:
Influenza, commonly known as "the flu", is an infectious disease caused by influenza viruses.

Influenza can contribute towards the development of pneumonia, sinus infections and worsening of previous health problems such as asthma or heart failure. Healthy people can get very sick from the flu and other respiratory viral infections and spread them to others. Therefore, early detection is essential for the effective management of these infections. Infection prevention and control measures including patient isolation, commencing anti-viral treatment and whether or not hospital admission is required can all be positively influenced by the rapid diagnosis of infection.

Current influenza testing can be performed by numerous methods. The gold standard is via molecular assays including rapid molecular assays and reverse transcription polymerase chain reaction (RT-PCR). Serological testing and antigen detection tests including immunofluorescence assays are other methods but the sensitivity and specificity for these tests are variable and tend to be lower than molecular testing methods.

In the United Kingdom (UK), influenza testing relies on clinical suspicion and the use of respiratory viral PCR in the laboratory. The turn-around-time for this can still take upto 48 hours. Point of care (POC) testing has been considered by Public Health England, as platforms with the potential to be used within 20 metres of patients and the results to be available within 10 to 90 minutes. This new device is a true point of care test which can be performed by the bedside with the results available within 10-15 mins.

This is a prospective single centre feasibility study carried out in an acute clinical setting, the Accident and Emergency (A+E) department of Imperial College Healthcare National Health Service (NHS) Trust (ICHNT).

The primary objective is to assess the feasibility of this novel single use product for the diagnosis of influenza and other respiratory pathogens in upper airway samples at the POC in acute clinical settings and compare the results against the conventional diagnostic methods of PCR testing in the laboratory and or rapid flu testing (Cepheid, Sunnyvale, CA, USA). While the secondary objective is to compare the results obtained in a clinical setting to the analytical study data and laboratory test on stored samples. A further objective is to develop a bank of research samples for further testing of the device in laboratory conditions. Sensitivity, specificity, positive predictive value and negative predictive value of the new POC device in fresh samples will be calculated and compared to the results on stored samples.

The patient will be seen in the clinical setting on a one off visit. Any adult presenting with Influenza Like Illness or a febrile illness associated with symptoms such as cough, sore throat or rhinorrhoea, and for whom a respiratory viral screen is clinically indicated will be recruited if they meet the eligibility criteria.

Consent will be taken by a qualified doctor, member of the local clinical care team, a research nurse or clinical fellow.

Participants will also be provided with contact details of the study co-ordination centre for future queries.

One nasal swab will be taken per patient recruited in addition to the swab(s) (nasal, nasopharyngeal or throat swab) taken for standard care. The routine screening sample(s) (Sample A) will be processed for standard PCR testing in the laboratory and/or rapid flu testing (Cepheid, Sunnyvale, CA, USA) as per standard clinical screening. The test sample (Sample B) will be taken for evaluation under the study and either: (i) transferred to the new device buffer tube and promptly tested in a test device or (ii) if no device is available for prompt testing, the swab will be transferred to a viral storage/transport buffer tube as per standard procedures and frozen for long-term storage and testing at a later date.

The swab will be rotated up to 5 times and held in place for 5-10 seconds. The swab will then be inserted into the single-use elution buffer tube containing the elution buffer and stirred 5 times. The swab will then be safely discarded in clinical waste. A volume of 200ul of buffer will then be transferred to the sample chamber of the device using the fixed volume pipette provided. The assay will be performed according to the 'Instructions for Use' provided with the device. Results require no calibration, interpretation, or calculation. The total time to result is expected to be approximately 10 minutes. The pathogens which will be tested in the test device include one or more of the following: influenza A, influenza B, respiratory syncytial virus, human rhinovirus/enterovirus, human metapneumovirus and parainfluenza viruses.

All tests performed on the device will be performed 'blinded', i.e. the operator will be unaware of the diagnostic standard of care result to ensure reading of results are not based upon results obtained with standard tests. The test result will not be disclosed to either the patient or the clinician. Each patient will be expected to participate for a total of 30 minutes.

As this is a feasibility study, diagnostic standard of care tests will be performed as per the clinical pathway with routine sample(s) (A) and the results of the test devices will not affect clinical decisions.

A minimum of 50 devices will be tested with fresh patient samples in a real life clinical setting. Opportunistic patient samples will be collected and banked throughout the study period. The aim will be to recruit as many patients as possible. A target of 200 patients has been set based on 1600 viral PCRs taken at ICHNT last year over the influenza period and a realistic estimate was made for the sample size for patients who may be willing to participate in the study presenting with Influenza Like Illness, with consideration of time and resource constraints. This data will be analysed to review the feasibility of this new device.

Medical and demographic data will be collected during the study and documented on the following case report forms (CRFs).

* Baseline CRF - Including demographic information, medical history, symptoms, signs and observations at the time of recruitment
* Results CRF - Including results from the POC device, how many devices were required to obtain a results, any issues with the device, results of the standard viral PCR results, patient outcomes and use of anti-viral treatment.

Additional data will be collected where required using the following CRFs:

* Adverse Events/Serious Adverse Events CRF.
* Withdrawal CRF - to be completed if patient withdraws consent. This data will be collected by a clinical research fellow or research nurses using participant hospital records or from the participant directly. In addition, pseudo-anonymised test results and imaging reports maybe collected. This could include but will not be limited to X-ray reports, CT scan reports, and pathology reports.

ELIGIBILITY:
Inclusion Criteria:

Any adult ≥18 years of age presenting to the A+E department with ILI or a febrile illness associated with symptoms such as cough, sore throat or rhinorrhoea, and for whom a respiratory viral screen is clinically indicated and who is:

* Able to provide written informed consent, or written informed assent by a relative or carer
* Recruited during initial medical assessment
* Able to comply with the study protocol

Exclusion Criteria:

* Previously recruited within 28 days of the current admission
* Enrolment in a trial of antimicrobial therapy
* If patients are unable to understand verbal or written information in English, hospital translation services will be sought but not guaranteed. However, if the team member seeking consent is not satisfied that the potential recruits' English language ability is sufficient to completely understand the study protocol and requirements (despite use of hospital translation services) then they will not be recruited to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any consenting adult presenting to the Accident and Emergency department with influenza like illness or a febrile illness associated with symptoms such as cough, sore throat or rhinorrhoea, and for whom a respiratory viral screen is clinically indicated will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Muir, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Suspected Influenza or Other Respiratory Viral Infection.: Any adult presenting to the Accident & Emergency department with influenza like illness or a febrile illness associated with symptoms such as cough, sore throat or rhinorrhoea, and for whom a respiratory viral screen is clinically indicated.
  For the purposes of this study one nasal swab will be taken from consenting adults.
  Point of care testing of respiratory viruses.: Single use point of care diagnostic device.
Period: Overall Study
Arm/Group | Suspected Influenza or Other Respiratory Viral Infection.
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Suspected Influenza or Other Respiratory Viral Infection.
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6

OUTCOME MEASURES:

1. Primary Outcome: Assessing the Feasibility of a Single Use Diagnostic Point of Care Test Against Standard Care Testing Methods, in a Real-life Clinical Setting.
Description: The primary outcome will be to review the feasibility and the diagnostic accuracy for viral respiratory pathogens in this novel device using fresh patients' samples in a real-life clinical setting compared to the standard diagnostic testing of a respiratory viral PCR in the laboratory and/or rapid flu swab (Cepheid, Sunnyvale, CA, USA) using sensitivity, specificity, positive predictive value and negative predictive values. A minimum of 50 devices will be tested with fresh patient samples in a real life clinical setting.
Time Frame: through study completion, an average of 1.5 years
Population: study terminated before results
Arm/Group | Suspected Influenza or Other Respiratory Viral Infection.
Number analyzed (Participants) | 0

2. Secondary Outcome: To Compare the Results Obtained in a Clinical Setting to the Analytical Study Data and Laboratory Tests on Stored Samples.
Description: The secondary outcome will be to review the feasibility and the diagnostic accuracy for viral respiratory pathogens in this novel device using patients' stored samples in a laboratory setting compared to the standard diagnostic testing of a respiratory viral PCR in the laboratory and/or rapid flu swab (Cepheid, Sunnyvale, CA, USA) using sensitivity, specificity, positive predictive value and negative predictive values.
Time Frame: through study completion, an average of 1.5 years
Population: outcome measure data not collected
Arm/Group | Suspected Influenza or Other Respiratory Viral Infection.
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Suspected Influenza or Other Respiratory Viral Infection.
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/50/NCT04431050/Prot_SAP_000.pdf